CLINICAL TRIAL: NCT02560922
Title: Pain Coping Skills Training for African Americans With Osteoarthritis
Acronym: STAART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-1189; AD-1408-19519 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2015-09-22; First posted 2015-09-25 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2018-05

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Knee Osteoarthritis; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pain Coping Skills Training (Experimental): This group will take part in an 11-week pain coping skills training (CST) intervention.
  Interventions: Behavioral: Pain Coping Skills Training (CST)
- Wait list Control (No Intervention): The other group will be the wait list group and will receive the pain CST program after completing all follow-up study measures.

INTERVENTIONS:
Behavioral: Pain Coping Skills Training (CST) — The pain CST intervention includes 11 individual sessions with a study counselor, delivered via telephone to enhance access and reach. The sessions include the following: general information about why pain coping skills training is important, training in specific pain coping skills (such as progressive muscle relaxation, communication, imagery, and activity pacing), and guided practice with each skill. The CST program will also include information about other behaviors important for OA, such as physical activity and weight management.
  Arms: Pain Coping Skills Training

SUMMARY:
This study will examine the effectiveness of an 11-session, culturally enhanced, telephone-based pain coping skills training program among African Americans with hip or knee osteoarthritis (OA). The study team will enroll n=248 African Americans with hip or knee OA. The participants will be randomized into two groups. One group will take part in an 11-week pain CST intervention. The other group will be a "wait list" that receives the pain CST program after completing all follow-up study measures. All study participants will be able to continue any other usual medical care for their OA during the study period. The pain CST intervention includes 11 individual sessions with a study counselor, delivered via telephone to enhance access and reach. The sessions include the following: general information about why pain coping skills training is important, training in specific pain coping skills (such as progressive muscle relaxation, communication, imagery, and activity pacing), and guided practice with each skill. The CST program will also include information about other behaviors important for OA, such as physical activity and weight management. The main study outcome will be the pain subscale of the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC). Other outcomes will include the WOMAC function subscale, Coping Strategies Questionnaire, Arthritis Self Efficacy Scale, depressive symptoms, Health-Related Quality of Life, and Patient Global Impression of Change.

DETAILED DESCRIPTION:
Background and Significance: OA is a leading cause of pain and disability. African Americans have a greater burden of OA. In this demographic group OA is more common and associated with more severe pain and activity limitations, compared with Caucasians. Prior research suggests that a program called pain Coping Skills Training (CST) has strong potential for helping African Americans with OA to reduce their symptoms. However, there are still some important limitations to what is known in this research, which limits putting this program into practice. First, there is a need to incorporate the perspectives of African Americans with OA, as well as other key Stakeholders, into this program. This is important for ensuring the program is culturally relevant and can be successfully used in a variety of clinical and community settings. Second, there is still a need for a study that will test the effectiveness of pain CST specifically among African Americans with OA in "real world" settings. Therefore the objective of this project is to examine the effectiveness of a culturally enhanced pain CST program among African Americans with OA.

Study Aims: This project has three specific aims: 1.) Engage African American patients with OA, their support partners, health care providers, clinic administrators, and public health representatives in a process of evaluating and enhancing a pain CST program for culturally appropriate content and dissemination potential. 2.) Examine the effectiveness of a 12-session, culturally enhanced, telephone-based pain CST program among African Americans with hip or knee OA. 3.) Examine whether individual patient characteristics are associated with different levels of improvement in the CST program. The long-term objective of this research is to develop and disseminate an evidence-based pain CST intervention among African Americans with OA, to reduce disparities in outcomes.

Study Description: Following the incorporation of Stakeholder perspectives into the pain CST program, the investigators will conduct a randomized controlled trial. The investigators will enroll n=248 African Americans with hip or knee OA. They will be randomized into two groups. One group will take part in a 2-week pain CST intervention. The other group will be a "wait list" that receives the pain CST program after completing all follow-up study measures. All study participants will be able to continue any other usual medical care for their OA during the study period. The pain CST intervention includes 12 individual sessions with a study counselor, delivered via telephone to enhance access and reach. The sessions include the following: general information about why pain coping skills training is important, training in specific pain coping skills (such as progressive muscle relaxation, communication, imagery, and activity pacing), and guided practice with each skill. The CST program will also include information about other behaviors important for OA, such as physical activity and weight management. The main study outcome will be the pain subscale of the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC). Other outcomes will include the WOMAC function subscale, Coping Strategies Questionnaire, Arthritis Self Efficacy Scale, depressive symptoms, Health-Related Quality of Life, and Patient Global Impression of Change. These measures were selected based on Stakeholder input and prior research that showed these outcomes are important to patients with OA. Statistical models will be used to compare outcomes between the two study groups at each time point: baseline, 12 weeks (after completion of the initial CST intervention), and 36 weeks (about 6 months after intervention completion). The investigators will also assess whether there are different levels of improvement in outcomes of the CST intervention, based on participant characteristics.

ELIGIBILITY:
Inclusion Criteria:

* African American (based on self-reported race)
* Diagnosis of hip or knee osteoarthritis; current joint symptoms

Exclusion Criteria:

* Diagnosis of gout (in knee or hip), rheumatoid arthritis, fibromyalgia, other systemic rheumatic disease
* Dementia or other memory loss condition
* Active diagnosis of psychosis, serious personality disorder, or current uncontrolled substance abuse
* Total hip / knee replacement surgery, other knee / hip surgery, anterior cruciate ligament tear, or other significant hip / knee injury in the past 6 months
* Severely impaired hearing or speech (patients must be able to participate in video-conference sessions)
* Unable to speak English
* Participating in another OA intervention or CST study
* Unwilling to be randomized either study arm
* Lower extremity paralysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2016-04; Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli D Allen, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Thurston Arthritis Research Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Dharmasri CJ, Griesemer I, Arbeeva L, Campbell LC, Cene CW, Keefe FJ, Oddone EZ, Somers TJ, Allen KD. Acceptability of telephone-based pain coping skills training among African Americans with osteoarthritis enrolled in a randomized controlled trial: a mixed methods analysis. BMC Musculoskelet Disord. 2020 Aug 14;21(1):545. doi: 10.1186/s12891-020-03578-7. PMID 32795282
- [Derived] Allen KD, Arbeeva L, Cene CW, Coffman CJ, Grimm KF, Haley E, Keefe FJ, Nagle CT, Oddone EZ, Somers TJ, Watkins Y, Campbell LC. Pain coping skills training for African Americans with osteoarthritis study: baseline participant characteristics and comparison to prior studies. BMC Musculoskelet Disord. 2018 Sep 19;19(1):337. doi: 10.1186/s12891-018-2249-6. PMID 30227841
- [Derived] Schrubbe LA, Ravyts SG, Benas BC, Campbell LC, Cene CW, Coffman CJ, Gunn AH, Keefe FJ, Nagle CT, Oddone EZ, Somers TJ, Stanwyck CL, Taylor SS, Allen KD. Pain coping skills training for African Americans with osteoarthritis (STAART): study protocol of a randomized controlled trial. BMC Musculoskelet Disord. 2016 Aug 23;17(1):359. doi: 10.1186/s12891-016-1217-2. PMID 27553385

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pain Coping Skills Training | Wait List Control
Started | 124 | 124
Completed | 98 | 112
Not Completed | 26 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Coping Skills Training | Wait List Control | Total
Number analyzed (Participants) | 124 | 124 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.8) | 58.9 (10.9) | 59.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 61 | 122
  Male | 63 | 63 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 116 | 116 | 232
  Unknown or Not Reported | 5 | 4 | 9
Some education above high school [Count of Participants; unit: Participants] | 92 | 95 | 187
Working [Count of Participants; unit: Participants] | 43 | 43 | 86
Married or living with partner [Count of Participants; unit: Participants] | 51 | 52 | 103
Low Perceived Income [Count of Participants; unit: Participants] — Self-report of either "just meet basic expenses" or "don't even have enough to meet basic expenses"
  Participants | 48 | 35 | 83
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 35.6 (8.4) | 34.8 (7.9) | 35.2 (8.2)
Number of Self-Reported Comorbidities [Mean (Standard Deviation); unit: comorbidities] | 8.2 (3.9) | 8.8 (4.0) | 8.5 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 3 and Change From Baseline to 9 Month in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Pain Subscale
Description: Change over time in the primary outcome measure for this study, the Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Pain Subscale is a measure of lower extremity pain. It includes 5 items rated on a Likert scale of 0 (no symptoms) to 4 (extreme symptoms), with a total range of 0-20 with higher scores indicating worse symptoms and function.
Time Frame: Baseline, 3 months and 9 months
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pain Coping Skills Training | Wait List Control
Number analyzed (Participants) | 124 | 124
units on a scale
  Baseline to 3 month change | -1.59 [-2.21 to -0.97] | -0.96 [-1.56 to -0.35]
  Baseline to 9 month change | -2.24 [-2.91 to -1.56] | -1.40 [-2.04 to -0.77]
Statistical Analysis 1: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 3 months; Test type: Superiority; p = 0.128, Mixed Models Analysis; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.45 to 0.18]
Statistical Analysis 2: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 9 months; Test type: Superiority; p = 0.068, Mixed Models Analysis; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.73 to 0.06]

2. Secondary Outcome: Change From Baseline to Month 3 and Change From Baseline to 9 Month in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Total Score
Description: In addition to the pain subscale, the WOMAC includes stiffness (2 items) and function (17 items) subscales. All items are listed rated on a Likert scale of 0 (no symptoms) to 4 (extreme symptoms), with ranges of 0-96 for the total score (pain, stiffness, and function subscales), with higher scores indicating worse symptoms and function.
Time Frame: Baseline, 3 months and 9 months
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pain Coping Skills Training | Wait List Control
Number analyzed (Participants) | 124 | 124
units on a scale
  Baseline to 3 month change | -6.60 [-9.10 to -4.10] | -3.98 [-6.42 to -1.55]
  Baseline to 9 month change | -8.81 [-11.58 to -6.05] | -5.50 [-8.11 to -2.89]
Statistical Analysis 1: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 3 months; Test type: Superiority; p = 0.129, Mixed Models Analysis; Mean Difference (Final Values) = -2.62, 95% CI 2-sided [-6.01 to 0.77]
Statistical Analysis 2: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 9 months; Test type: Superiority; p = 0.084, Mixed Models Analysis; Mean Difference (Final Values) = -3.31, 95% CI 2-sided [-7.07 to 0.44]

3. Secondary Outcome: Change From Baseline to Month 3 and Change From Baseline to 9 Month in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Function Subscale
Description: In addition to the pain subscale, the WOMAC includes stiffness (2 items) and function (17 items) subscales. All items are listed rated on a Likert scale of 0 (no symptoms) to 4 (extreme symptoms), with ranges of 0-68 for the function subscale, with higher scores indicating worse symptoms and function.
Time Frame: Baseline, 3 months and 9 months
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pain Coping Skills Training | Wait List Control
Number analyzed (Participants) | 124 | 124
units on a scale
  Baseline to 3 month change | -4.08 [-5.93 to -2.22] | -2.46 [-4.27 to -0.65]
  Baseline to 9 month change | -5.60 [-7.69 to -3.51] | -3.41 [-5.39 to -1.43]
Statistical Analysis 1: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 3 months; Test type: Superiority; p = 0.209, Mixed Models Analysis; Mean Difference (Final Values) = -1.61, 95% CI 2-sided [-4.14 to 0.91]
Statistical Analysis 2: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 9 months; Test type: Superiority; p = 0.128, Mixed Models Analysis; Mean Difference (Final Values) = -2.20, 95% CI 2-sided [-5.03 to 0.63]

4. Secondary Outcome: Change From Baseline to Month 3 and Change From Baseline to 9 Month in PROMIS Pain Interference (Short Form 6a)
Description: The PROMIS Pain Interference (Short Form 6a) instrument measures the self-reported consequences of pain across aspects of life including social, cognitive, emotional, physical and recreational activities; this instrument refers to the past seven days. This validated scale has five response options, with scores ranging from one to five. Scores are converted to t-scores, and higher scores indicate greater pain interference.
Time Frame: Baseline, 3 months and 9 months
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: t-score
Arm/Group | Pain Coping Skills Training | Wait List Control
Number analyzed (Participants) | 124 | 124
t-score
  Baseline to 3 month change in t-score | -2.63 [-3.66 to -1.60] | -1.80 [-2.80 to -0.80]
  Baseline to 9 month change in t-score | -2.75 [-3.83 to -1.67] | -1.61 [-2.63 to -0.60]
Statistical Analysis 1: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 3 months; Test type: Superiority; p = 0.222, Mixed Models Analysis; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-2.18 to 0.51]
Statistical Analysis 2: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 9 months; Test type: Superiority; p = 0.128, Mixed Models Analysis; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-2.60 to 0.33]

5. Secondary Outcome: Change From Baseline to Month 3 and Change From Baseline to 9 Month in Short Form (SF)-12 Physical Component Health Score
Description: This 12-item measure covers domains of general health, physical health, work and activity limitations, and emotional health. Mental Health and Physical Health Composite Scores were computed, both of which range from 0-100 with lower scores indicating poorer health.
Time Frame: Baseline, 3 months and 9 months
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pain Coping Skills Training | Wait List Control
Number analyzed (Participants) | 124 | 124
units on a scale
  Baseline to 3 month change | 2.60 [1.05 to 4.15] | 0.89 [-0.63 to 2.40]
  Baseline to 9 month change | 2.47 [0.86 to 4.08] | 1.74 [0.21 to 3.26]
Statistical Analysis 1: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 3 months; Test type: Superiority; p = 0.111, Mixed Models Analysis; Mean Difference (Final Values) = 1.71, 95% CI 2-sided [-0.40 to 3.82]
Statistical Analysis 2: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 9 months; Test type: Superiority; p = 0.502, Mixed Models Analysis; Mean Difference (Final Values) = 0.73, 95% CI 2-sided [-1.42 to 2.88]

6. Secondary Outcome: Change From Baseline to Month 3 and Change From Baseline to 9 Month in SF-12 Mental Component Health Score
Description: as for outcome 5
Time Frame: Baseline, 3 months and 9 months
Population: This variable was analyzed as a change score (baseline to 3-month and baseline to 9-month), due to normality assumptions. Therefore only participants with complete data at baseline and follow-up could be included in the analysis, resulting in a smaller sample than the total population.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pain Coping Skills Training | Wait List Control
Number analyzed (Participants) | 117 | 112
units on a scale
  Baseline to 3 month change | -0.72 [-2.08 to 0.64] | -1.48 [-2.82 to -0.15]
  Baseline to 9 month change | -0.57 [-2.13 to 0.99] | -2.28 [-3.77 to -0.79]
Statistical Analysis 1: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 3 months; Test type: Superiority; p = 0.433, Mixed Models Analysis; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-1.15 to 2.66]
Statistical Analysis 2: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 9 months; Test type: Superiority; p = 0.120, Mixed Models Analysis; Mean Difference (Final Values) = 1.71, 95% CI 2-sided [-0.45 to 3.86]

7. Secondary Outcome: Change From Baseline to Month 3 and Change From Baseline to 9 Month in Coping Strategies Questionnaire (CSQ)
Description: This scale includes 48 items that assess 6 cognitive domains (Catastrophizing, Diverting Attention, Ignoring Sensations, Coping Self-Statements, Reinterpreting Pain Sensations, Praying-Hoping) and 1 behavioral domain (Increasing Behavioral Activities). Each domain includes 6 items, and participants rate the frequency of their use of specific coping strategies on a 7-point Likert scale from 0 ("Never do that") to 6 ("Always do that"). A Total Coping Attempts score was created, which includes 5 cognitive domains and 1 behavioral domain but excludes the Catastrophizing domain, similar to prior studies. Total range is 252, with higher scores indicating more coping attempts.
Time Frame: Baseline, 3 months, 9 months
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pain Coping Skills Training | Wait List Control
Number analyzed (Participants) | 124 | 124
units on a scale
  Baseline to 3 month change | 16.46 [11.68 to 21.25] | 1.15 [-3.52 to 5.83]
  Baseline to 9 month change | 9.27 [4.26 to 14.28] | -2.40 [-7.18 to 2.37]
Statistical Analysis 1: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 3 months; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 15.31, 95% CI 2-sided [9.09 to 21.53]
Statistical Analysis 2: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 9 months; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 11.67, 95% CI 2-sided [5.08 to 18.27]

8. Secondary Outcome: Change From Baseline to Month 3 and Change From Baseline to 9 Month in Patient Health Questionnaire 8 (PHQ-8)
Description: This 8-item survey of depressive symptoms includes items corresponding to the depression criteria listed in the Diagnostic and Statistics Manual Fourth Edition (DSM-IV) [38]. All items are scored as 0 (not at all) to 3 (nearly every day), with higher scores indicating more depressive symptoms.
Time Frame: Baseline, 3 months and 9 months
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pain Coping Skills Training | Wait List Control
Number analyzed (Participants) | 124 | 124
units on a scale
  Baseline to 3 month change | -0.32 [-1.12 to 0.48] | 0.18 [-0.59 to 0.96]
  Baseline to 9 month change | -0.89 [-1.78 to 0] | 0.13 [-0.71 to 0.97]
Statistical Analysis 1: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 3 months; Test type: Superiority; p = 0.356, Mixed Models Analysis; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.57 to 0.57]
Statistical Analysis 2: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 9 months; Test type: Superiority; p = 0.087, Mixed Models Analysis; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-2.19 to 0.15]

9. Secondary Outcome: Change From Baseline to Month 3 and Change From Baseline to 9 Month in Arthritis Self-Efficacy Scale
Description: This scale includes 8 items asking respondents how certain they are that they can manage arthritis pain and keep it from interfering with specific activities All items are scored on a scale of 1 (very uncertain) to 10 (very certain), with higher scores indicating greater self-efficacy for managing arthritis symptoms.
Time Frame: Baseline, 3 months and 9 months
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pain Coping Skills Training | Wait List Control
Number analyzed (Participants) | 124 | 124
units on a scale
  Baseline to 3 month change | 0.81 [0.50 to 1.11] | -0.20 [-0.50 to 0.09]
  Baseline to 9 month change | 0.46 [0.14 to 0.78] | -0.21 [-0.51 to 0.10]
Statistical Analysis 1: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 3 months; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [0.61 to 1.41]
Statistical Analysis 2: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between group difference in change from baseline to 9 months; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [0.24 to 1.09]

10. Secondary Outcome: Patient Global Impression of Arthritis Symptom Change From Baseline (BL) at 3 and 9 Months
Description: This measure asks participants to describe their change in pain on a 7-point rating scale with the following options: "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," and "very much worse." The total range is 0-7, with lower scores indicating more improvement.
Time Frame: Baseline, 3 months and 9 months
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pain Coping Skills Training | Wait List Control
Number analyzed (Participants) | 124 | 124
units on a scale
  Self reported change in symptoms between BL and 3m | 2.91 [2.67 to 3.14] | 4.18 [3.95 to 4.40]
  Self reported change in symptoms between BL and 9m | 3.25 [2.99 to 3.52] | 4.13 [3.87 to 4.38]
Statistical Analysis 1: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between-group difference in self-reported change in symptoms (from baseline) at 3 months; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-1.60 to -0.95]
Statistical Analysis 2: Comparison: Pain Coping Skills Training vs Wait List Control; Test of between-group difference in self-reported change in symptoms (from baseline) at 9 months; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-1.24 to -0.51]

ADVERSE EVENTS:
Time Frame: Data were collected for 12 months, ending at participants' final follow up time point.
Arm/Group | Pain Coping Skills Training | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/124
Serious Adverse Events (participants affected / at risk) | 15/124 | 6/124
Other Adverse Events (participants affected / at risk) | 0/124 | 0/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pain Coping Skills Training (N=124) | Wait List Control (N=124)
lower GI bleed (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest Pain (Cardiac disorders) | 2 (2) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 2 (2) | 0 (0)
Total knee arthroplasty of right knee (Surgical and medical procedures) | 1 (1) | 0 (0)
Laparoscopic Gastrocutaneous Fistula Takedown (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical removal of lymphedema lobe on left leg (Surgical and medical procedures) | 1 (1) | 0 (0)
Accidental exposure to trichoroacetic acid (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Food impaction in esophagus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured ribs (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia and dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Implantation of catheter-delivered aortic heart valve, insertion of temporary pacemaker, introductio (Surgical and medical procedures) | 1 (1) | 0 (0)
Sepsis 2/2 Abdominal cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT02560922/Prot_SAP_000.pdf